CLINICAL TRIAL: NCT03176342
Title: Drug Patch Tests, Enzyme-linked Immunosorbent Spot Assay (Elispot) and Lymphocyte Transformation Tests in Patients With Severe Cutaneous Adverse Reaction to Drugs (SCARs)
Brief Title: Drug Patch Tests in Patients With Severe Cutaneous Adverse Reaction to Drugs (SCARs)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pawinee Rerknimitr, Assistant professor, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 204/59
Record Dates: First submitted 2017-06-02; First posted 2017-06-05 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Drug Reaction
Keywords: Drug patch tests
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Patch Tests; Enzyme-Linked Immunospot Assay

STUDY DESIGN:
Oversight: FDA-regulated Drug: No

ARMS (1):
- patch test arm (Experimental): Patch test by selected allergens and drawing blood for ELIspot and LTT
  Interventions: Other: patch test

INTERVENTIONS:
Other: patch test — Patch test allergen from chemotechnique diagnostics, pure drug and drug as is combine with petrolatum or aqueous.
  Other Names: Enzyme-linked immunosorbent spot assay (ELIspot) and lymphocyte transformation test (LTT)

SUMMARY:
The study is about drug patch tests in patients who have history of severe cutaneous drug reaction including Steven Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), Drug-induced eosinophilia and systemic symptoms (DRESS), AGEP (Acute generalized exanthematous pustulosis) and generalized bullous fixed drug eruptions. This study also investigate in Enzyme-linked immunosorbent spot assay (ELIspot) and lymphocyte transformation test. We also trying to prove the correlation among result of drug patch tests, ELIspot and LTT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of Steven Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), drug-induced eosinophilia and systemic symptoms (DRESS), acute generalized exanthematous pustulosis (AGEP), generalized bullous fixed drug eruption in the past 24 months.
* Age more than 18 years old

Exclusion Criteria:

* Receiving immunosuppressive drugs or more than 10 mg/day of prednisolone within 1 month.
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08-04 (Actual); Primary Completion 2017-08-03 (Estimated); Study Completion 2017-08-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of positive drug patch test results. | 3 years

SECONDARY OUTCOMES:
correlation of drug patch test results, ELIspot and lymphocyte transformation test. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Dermatology, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand